CLINICAL TRIAL: NCT03361618
Title: Effect of Oral Zinc Sulfate Supplementation on Enzymes of Urate Pathway in Spermatozoa and Seminal Plasma of Iraqi Asthenospermic Patients
Brief Title: Effect of Oral Zinc Sulfate Supplementation on Enzymes of Urate Pathway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babylon University (Other)
Collaborators: Ministry of Health, Iraq (Network)
Responsible Party: Principal Investigator, mahmoud hussein hadwan, Principal Investigator Dr. Mahmoud Hussein Hadwan, Babylon University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Babil-5
Record Dates: First submitted 2017-11-07; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Infertility Unexplained
Keywords: Uric acid; Adenosine deaminase; Zinc Sulfate; 5'-nucleotidase; Asthenospermia.; Xanthine oxidase
MeSH Terms: conditions — Asthenozoospermia | interventions — Zinc Sulfate

STUDY DESIGN:
Intervention Model Description: Semen volume after treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zinc sulfate (Experimental): 60 subfertile (age 32.5±3.23 year) men with asthenozoospermia was treated with zinc sulfate, every participant took two capsules of zinc sulfate per day for three months (each one 220 mg).
  Interventions: Dietary Supplement: Zinc Sulfate
- Healthy control (No Intervention): 60 fertile (age 31.6±3.3 year) men, no treatment.

INTERVENTIONS:
Dietary Supplement: Zinc Sulfate — The subfertile group treated with zinc sulfate, every participant took two capsules of zinc sulfate per day for three months (each one 220 mg).
  Arms: Zinc sulfate

SUMMARY:
Although many reports have investigated the relationship between subfertility and uric acid levels in semen, to the best of author knowledge, there is no study have been published to yet focus on the effects of asthenospermia treatments, such as given an oral zinc supplementation, on the activity of urate-related enzymes, which are important in fertility of human.

DETAILED DESCRIPTION:
The present study was designed to investigate the effect of zinc supplementation on the qualitative and quantitative characteristics of semen, along with uric acid levels and urate-related enzymes in the seminal plasma and spermatozoa of asthenospermic males.

ELIGIBILITY:
Inclusion Criteria:

* The presence of asthenozoospermia in the semen sample.
* Must be unable to reproduce.

Exclusion Criteria:

* the absence of endocrinopathy, varicocele, and female factor infertility. Smokers and alcoholic men were excluded from the study because of their recognized high seminal ROS levels and decreased antioxidant levels.

Ages: 26 Years to 36 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male that undergo the presence of asthenozoospermia in the semen sample.
Enrollment: 120 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2012-06-01 (Actual); Study Completion 2012-06-01 (Actual)

PRIMARY OUTCOMES:
Measurement the uric acid level in spermatozoa and seminal plasma by using spectrophotometer. | up to three months.
  Clinical parameter

SECONDARY OUTCOMES:
Measurement the adenosine deaminase activity in spermatozoa and seminal plasma by using spectrophotometer. | up to three months.
  Enzyme
Measurement the xanthine oxidase activity in spermatozoa and seminal plasma by using spectrophotometer. | up to three months.
  Enzyme
Measurement the 5'-nucleotidase activity in spermatozoa and seminal plasmaby using the spectrophotometer. | up to three months.
  Enzyme

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Razzaq A. Alsalman, PhD, Study Chair — University of Babyblon; Lamia A. Almashhedy, PhD, Study Director — University of Babyblon; Mahmoud Hussein Hadwan, PhD, Principal Investigator — University of Babyblon; Abdulsamie H Alta'ee, PhD, Study Director — University of Babyblon
Locations (1):
- Mahmoud Hussein Hadwan, Hillah, Babylon, Iraq

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Alsalman ARS, Almashhedy LA, Alta'ee AH, Hadwan MH. Effect of Zinc Supplementation on Urate Pathway Enzymes in Spermatozoa and Seminal Plasma of Iraqi Asthenozoospermic Patients: A Randomized Controlled Trial. Int J Fertil Steril. 2020 Jan;13(4):315-323. doi: 10.22074/ijfs.2020.5760. Epub 2019 Nov 11. PMID 31710193